CLINICAL TRIAL: NCT03246880
Title: Clinical Trial To Evaluate the Efficacy and Safety of CKD-397 in Benign Prostatic Hyperplasia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 150BPH15018
Record Dates: First submitted 2015-09-02; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Tamsulosin 0.2mg+Tadalafil 5mg (Experimental): Tamsulosin 0.2mg+Tadalafil 5mg, po, q.d.
  Interventions: Drug: Tamsulosin 0.2mg; Drug: Tadalafil 5mg
- Tamsulosin 0.2mg (Active Comparator): Tamsulosin 0.2mg, po, q.d.
  Interventions: Drug: Tamsulosin 0.2mg
- Tadalafil 5mg (Active Comparator): Tadalafil 5mg, po, q.d.
  Interventions: Drug: Tadalafil 5mg

INTERVENTIONS:
Drug: Tamsulosin 0.2mg — per oral for 12weeks after 2~4weeks run-in period
  Arms: Tamsulosin 0.2mg; Tamsulosin 0.2mg+Tadalafil 5mg
Drug: Tadalafil 5mg — per oral for 12weeks after 2~4weeks run-in period
  Arms: Tadalafil 5mg; Tamsulosin 0.2mg+Tadalafil 5mg

SUMMARY:
A Multicenter, Randomized, Double-blind, Active-controlled, Parallel group, Phase III Clinical Trial To Evaluate the Efficacy and Safety of CKD-397 in Benign Prostatic Hyperplasia Patients.

ELIGIBILITY:
Inclusion Criteria:

[Visit 1]

1. Male Aged of 45 or above
2. Patients must have a diagnosis of Benign Prostatic Hyperplasia
3. IPSS(International Prostate Symptom Score) questionnaire total score ≥ 13
4. Signed and dated informed consent document indicating that the patient

[Visit 2]

1. IPSS(International Prostate Symptom Score) questionnaire total score ≥ 13
2. 15mL/s ≥ Qmax ≥ 4mL/s, if voided volume ≥ 120ml
3. PVR(post-void residual urine volume) ≤ 250ml

Exclusion Criteria:

1. Patients have ever taken Finasteride in 3 months or Dutasteride in 6 months
2. Patients with prostate cancer or PSA > 10ng/ml
3. Patients with other disease which could have influence on urine flow rate except BPH(benign prostatic hyperplasia )
4. Patients with a history of operation on prostate which could have influence on the result and need to have surgery.
5. Patients with acute urinary retention in 3months
6. Patients with a history of drug or alcohol abuse within 6 months
7. Patients have cardiovascular disease or associated disease which is not controlled.
8. Patients who need to take Nitrates, alpha blocker, Nitric Oxide Donor
9. Patients with orthostatic hypotension
10. Patients with a history micturition syncope
11. Patients with severe or malignant retinopathy
12. Patients have a visual disturbance by Non-arteritic anterior ischemic optic neuropathy
13. Patients with a congestive disease like galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
14. Serum creatinine > upper Normal Limit*2, AST/ALT > upper Normal Limit*3
15. Patient with uncontrolled diabetes(HbA1C>9%)
16. Patients have a history of malignant tumor within 5 years
17. Patients have hypersensitivity reaction on this drug.
18. Patients treated with other investigational product within 4 weeks at first time taking the investigational product
19. Not eligible to participate for the study at the discretion of investigator

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The mean change of the total score on IPSS questionnaire(International Prostate Symptom Score ) | From baseline at week 12

SECONDARY OUTCOMES:
The mean change of scores on three questionnaire, Qmax(maximum flow rate(urine), PVR(post-void residual urine volume) | From baseline at week 12
  IPSS questionnaire(International Prostate Symptom Score ), IIEF-5(International Index of Erectile Function-5) questionnaire Change in score, ICIQ-MLUTS(International Consultation on Incontinence Modular Questionnaire-Male Lower Urinary Tract Symptoms) questionnaire Change in score
The mean change of scores on IPSS ( International Prostate Symptom Score ), ICIQ-MLUTS( International Consultation on Incontinence Modular Questionnaire-Male Lower Urinary Tract Symptoms) questionnaire Change in score | From baseline at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Soo Choo, M.D., Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea